### **INFORMED CONSENT FORM (ICF)**

# BRIDGING TRIAL TO EVALUATE THE INFECTIVITY EQUIVALENCE OF CURRENT AND NEW LOTS OF PLASMODIUM FALCIPARUM STRAIN NF54 (CLONE 3D7) WITHIN THE WRAIR CONTROLLED HUMAN MALARIA INFECTION (CHMI) MODEL

NCT# 03882528

**Document Date: 21FEB2019** 



#### DEPARTMENT OF THE ARMY

WALTER REED ARMY INSTITUTE OF RESEARCH 503 ROBERT GRANT AVENUE SILVER SPRING, MD 20910-7500

**WRAIR # 2572** 

Version 4, Date: <u>21FEB2019</u>

## Walter Reed Army Institute of Research Consent for Research Participation

**Title:** Bridging Trial to Evaluate the Infectivity Equivalence of Current and New Lots of Plasmodium falciparum strain NF54 (clone 3D7) within the WRAIR Controlled Human Malaria Infection (CHMI) Model

**Sponsor:** The Surgeon General, Department of the Army

**Funder:** Military Infectious Diseases Research Program (MIDRP)

Principal Investigator (PI): James E. Moon, MD Colonel, US Army, WRAIR

**Contact Info:** 301-319-9176 james.e.moon.mil@mail.mil

**IND Number:** 18495

You are being asked to take part in a research study. This study is supported by the United States Department of Defense. The box below tells you important things you should think about before deciding to join the study. We will provide more detailed information below the box. Please ask questions about any of the information before you decide whether to participate. You may also wish to talk to others (for example, your family, friends, or your doctor) about this study, before agreeing to join.

Please contact one of the below if you have any questions concerning the study or if you have any other questions or concerns.

James E. Moon, MD Colonel, US Army (301) 319-9176

WRAIR Clinical Trials Center \* (301) 319-9660

\*Open 6:00AM-2:30PM Monday-Friday

#### **Key Information for You to Consider**

- Voluntary Consent. You are being asked to volunteer for a research study. It is up to you whether you choose to participate or not. There are no penalties and you will not lose anything if you decide not to join or if after you join, you decide to quit. However, if you decide to leave the study after you have been challenged with malaria, you will be asked to complete follow-up visits, diagnostic tests for malaria, treatment, and safety blood work to ensure your safety.
- Purpose. We are doing this research to evaluate how well a certain batch
  of malaria parasites causes infection in humans. Up to 12 individuals will
  participate in this trial
- **Duration.** Your part of the study will last up to 12 weeks (approximately 3 months), including today's screening visit.
- Procedures and Activities. During this study we will ask you to undergo exposure to malaria infection through mosquito bites, and then be followed for approximately one month, during which time YOU ARE EXPECTED TO BECOME INFECTED WITH MALARIA. During most of this period you will have daily blood draws and visits with medical providers to monitor your safety and look for evidence of infection. If and when you are diagnosed with malaria you will be given effective treatment to cure it. During the part of the month when you are most likely to develop malaria, you will be asked to spend up to 10 nights in a local hotel.
- Risks. Most studies have some possible harms that could happen to you
  if you join. In this study, we expect that YOU WILL BECOME INFECTED
  WITH MALARIA, but you will monitored, and given effective treatment to
  cure your infection once it occurs. Other risks are described elsewhere in
  this document.
- **Benefits**. There is no direct benefit to you for participating in this study. There may be a general health benefit from getting examined by a doctor and having blood tests done for your general health. Others may benefit in the future from the information that will be learned from the study.
- Alternatives. Participation is voluntary and the only alternative is to not participate.

#### Why are we doing this research?

You are being asked to participate in a research study evaluating how well a certain batch of malaria parasites causes infection in humans.

The only way to prove new drugs and vaccines will protect humans against malaria is to give them to human subjects and then expose those subjects to malaria to see if they are protected. This exposure can be accomplished by sending the subjects to countries and environments where malaria is present (i.e., Africa, Asia, South America, etc.), or by purposefully exposing them to malaria in a controlled environment.

It is this second method we are evaluating in this trial. For over 30 years, researchers from the Department of Defense and other organizations worldwide have utilized controlled exposure to malaria, known as "malaria challenge" or "controlled human malaria infection (CHMI)" to safely evaluate how well new drugs and vaccines work in preventing malaria. In a typical CHMI, subjects are exposed to a known type of malaria parasite through the bites of a small number of infected mosquitoes, and then are followed for approximately 1 month to see if they develop symptoms or other signs of malaria infection. Subjects who are diagnosed with malaria during this time are treated. Those who do not develop malaria during this period are considered to have been protected from infection by whatever drug or vaccine was being tested.

The issue at hand is that the batch of malaria parasites we have used for CHMI for many years is running out. We have developed a new batch of the same parasites. However, before we can use these parasites in drug or vaccine trials we have to prove that they act just like the old batch of parasites, and can cause predictable malaria infection in humans. It is for this purpose that we are conducting the trial described in this document.

#### How long will I be in this research study?

If you complete the study, you will be in the study up to approximately 12 weeks (or about 3 months including screening period). A study schedule will be provided along with this form. It lists the study activities and gives the approximate length of time for each study visit.

#### Where will this study take place?

The screening visit(s) and malaria challenge will take place at the Walter Reed Army Institute of Research (WRAIR) in Silver Spring, Maryland. After the malaria challenge the location of the overnight stays or the "hotel phase" will be in a hotel close to WRAIR.

#### What will happen if I decide to be in this research study?

If you agree to be in this research, you will be expected to complete a number of visits and procedures, beginning with today's screening visit. A basic outline of these activities is as follows:

#### Screening Visit (up to 2 months before the malaria challenge day)

- Your first visit, which you can do today, is the screening visit. If you agree to be in this study, you will be asked to sign this consent form and an HIV test consent form. You must take a short quiz, to test your understanding of the study, and score at least 80%, or get 8 out of 10 correct. If you do not score 80% on your first try, we will review the study information with you, and you will be able to take the quiz again. If you get less than 80% the second try, you will not be able to be in the study.
- You will be able to speak with a study physician who will get your medical history, perform a physical examination, and answer any of your questions.

Version 4, Date: <u>21FEB2019</u>

You will give blood samples for laboratory tests. We will collect about 2 1/3 tablespoons (~35 mL) of blood by placing a small needle in a vein in your arm. The blood tests will include complete blood count (CBC), liver and kidney function tests, sickle cell test (a type of blood disorder), glucose (a type of sugar in your blood), and tests for HIV, hepatitis B and hepatitis C.

- An electrocardiogram or EKG (tracing of the electrical action in your heart) will be performed. This is a simple, painless test in which leads are attached to your chest, arms and legs. It shows us the "electrical activity" of the heart, and can reveal warning signs for heart disease.
- If you are a female, a urine pregnancy test will be performed.

If any of your test results are abnormal, you will be informed about the test result and instructed to see your primary care provider. If you are female and your pregnancy test is positive, you will not be able to be in the study. At your request, we will provide you a copy of your laboratory test results. State regulations require that if any of your tests show that you have HIV, hepatitis B, or hepatitis C infection, we must report the information to the Maryland Department of Health. If you are a military service member, this information will also be reported to the military preventive medicine service.

#### Malaria Challenge

The malaria challenge will take place at the Walter Reed Army Institute of Research Insectary, which is located in building 503 Robert Grant Avenue, Silver Spring, MD.

The malaria challenge will use mosquitoes that are raised in a laboratory. The malaria parasite used in the malaria challenge can be cured with medication.

During the malaria challenge, you will be asked to do the following:

- You must provide the names and phone numbers of at least 2 emergency contacts to the study staff, and agree that they can be contacted before the challenge.
- You will be asked to NOT use any cologne, perfume, after-shave lotion, deodorant soap or body creams/lotions on any part of your body because they may stop the mosquitoes from biting.
- We will collect about 2/3 tablespoon (~10 mL) of your blood for safety laboratory tests and a baseline test to show you did not have malaria before you were challenged.
- If you are a female, you will have a urine pregnancy test. If your pregnancy test is positive, we will not allow you to be bitten by infected mosquitoes.
- Five mosquitoes will be placed in the container and allowed to bite you through mesh for 5 minutes. If fewer than 5 malaria-infected mosquitoes bite you, more will be added to the container and allowed to bite you for another 5 minutes. We will do this until a total of 5 malaria-infected mosquitoes have bitten you.

- You will be asked to stay for at least 30 minutes after the challenge so we can monitor you for any reactions.
- You will be given a card that shows that you have been bitten by mosquitoes carrying malaria parasites. The card will have the contact information of the study principal investigator. You will be asked to carry this card with you at all times until the end of the study.
- In the days after the challenge, you will be checked for signs and symptoms of malaria infection. The expectation is that YOU WILL GET MALARIA FROM THE MOSQUITO BITES.
- You will be instructed to contact the study personnel immediately should you develop any signs and/or symptoms that may be consistent with malaria (as described in section 12).

#### Post-Malaria Challenge: (Day 1 to morning of Day 9 after the malaria challenge)

From Day 1 to Day 8 after challenge, you will be required to come to the clinic once a day for brief visits to have a small amount of blood drawn (< 1 teaspoonful, ~2 to 4 mL each time) to check for the presence of malaria in your blood. You will also be seen in the clinic on the morning of Day 9 after challenge for the same purpose. Though, the blood draw on this visit will be larger (~3.5 tablespoonsful, ~56 mL), as the study will be taking blood both to check for the presence of malaria and for future malaria research. While it is unlikely you will develop malaria this early, if a diagnosis is made, you will be treated.

#### Hotel Phase: (Evening of Day 9 to Day 19 after the malaria challenge)

Starting on the evening of Day 9 after the malaria challenge, you will be required to spend every night at a designated hotel for up to approximately 10 nights. During the day, you can leave the hotel to go to work, school, and your other regular activities.

The clinical team will be at the hotel at all times. During the post-malaria challenge hotel phase, expect the following:

- You must check in with study staff in the hotel each morning and each evening. Each morning you will be seen by a study doctor, and your blood will be drawn and tested for malaria parasites (< 1 teaspoonsful, ~2 to 4 mL each time). Each afternoon you must check in with study staff to report how you are feeling and determine if you should be seen again that day. If you develop symptoms of malaria, your blood may be drawn more frequently to determine if you have malaria.</p>
- A study doctor will be in the hotel at all times. If you work at night, the study staff will work with your schedule, but you will still need to sleep at the hotel.
- If the study doctor determines that you have malaria, you will be treated and will
  continue to have daily visits. You will be allowed to leave the hotel after you

complete the treatment and a study physician determines that it will be safe for you to do so.

- WRAIR will pay for the hotel room stay. You will have to pay for all of your other expenses such as long-distance phone calls, meals, movies ordered in your room, and any other expenses.
- Malaria symptoms may develop either before or after the parasites are seen in your blood.
- Symptoms of malaria may include fever, headache, joint aches, tiredness, body aches, shaking chills, nausea, diarrhea, low back pain, and sometimes stomach tenderness
- If you are diagnosed with malaria, an extra blood sample will be taken for safety labs to assess your wellbeing (~1/2 tablespoonsful, ~8 mL).
- If you are diagnosed with malaria, you will be treated with an FDA-approved drug for malaria. You will be seen by the clinical study team every day until you complete the treatment course.
- If you are diagnosed with malaria, blood samples will continue to be collected once a day (< 1 teaspoonful, ~2 to 4 mL each time) to make sure that malaria parasites are no longer in your blood. This is the best way for the study team to determine if the malaria treatment is working. These blood collections will end after you have no evidence of malaria parasites for 3 days.
- If you get malaria, finish the treatment, and the parasites can no longer be found in your blood, the study doctor may release you from the hotel and daily visits.
- If you have chest pain, difficulty breathing, palpitations, or any other complaints AT ANY TIME after the challenge, you must notify the study staff immediately, so we can determine whether you need to see our study physician.

#### Post-Challenge Follow-Up Visits:

You will be asked to return to the WRAIR CTC for several follow-up visits after the hotel phase.

- If you have not developed malaria by the morning of Day 19, you will be empirically (that is, without a diagnosis) treated for malaria, and will be required to return to WRAIR CTC for necessary daily visits until you have completed the necessary treatment and parasite clearance blood tests (< 1 teaspoonful, ~2 to 4 mL each time).
- If you have been diagnosed but not completed your treatment for malaria by the morning of Day 19, you will be required to return to WRAIR CTC for necessary daily visits until you have completed the necessary treatment and parasite clearance blood tests (< 1 teaspoonful, ~2 to 4 mL each time).

 Your last visit will take place at the WRAIR CTC on Day 28 (+/- 7 days). At this visit a final evaluation will be performed by a study physician, and blood collected for safety labs and future malaria research (~4 tablespoonsful, ~58 mL).

#### What requirements do I have to meet in order to participate in this study?

You may be allowed to participate in the study if you meet the following requirements:

- You are between the ages of 18 and 50 years old.
- You are willing and able to participate in all planned study visits for the duration of the study.
- You are in good general health based on your medical history, physical examination, EKG, and screening laboratories.
- You are able to understand and sign this informed consent.
- You pass the written test called the 'Assessment of Understanding' with a score of at least 80% (8 out of 10 questions correct).
- You agree not to donate blood during the study and for 3 years after the malaria challenge.
- You agree not to travel to place(s) where there is malaria during the time of the study.
- If you are a female, you must agree to consistently use effective birth control (e.g., oral or implanted contraceptives, intrauterine device (IUD), diaphragm with spermicide, abstinence, cervical cap) during the period from the day of screening (today) through 3 months after the malaria challenge.
- You must be willing to take anti-malarial treatment after CHMI, if indicated.
- You must agree to stay in a pre-determined hotel near the WRAIR during the designated post-CHMI follow-up period from approximately 9 days after malaria challenge until 19 days after challenge or antimalarial treatment is completed, whichever comes first.
- If you are a federal employee (military or civilian), you must have approval from your supervisory chain to participate. The appropriate approval form will be provided to you.

You are not allowed to participate in this study if any of the following criteria apply to you:

- Any history of malaria infection or having been given a malaria vaccine
- Any history of travel to a country with the type of malaria we are studying in the past 6 months, or planned travel to such an area during the course of the study

- Any history of having lived in an area with the type of malaria we are studying for more than 5 years.
- Any use of medications that prevent or treat malaria during the 1 month prior to challenge or planned use during the study (outside of the drugs provided by the study team).
- Any serious medical illness or condition involving the heart, liver, lungs, or kidneys
- Any significant risk for developing heart disease in the next 5 years. The risk for developing heart disease in the next 5 years will be determined by a combination of the following factors: high blood pressure, smoking, weight, family history of heart disease and the presence of diabetes
- Any medical illness or condition involving your blood or immune system (to include sickle cell trait or thalassemia trait)
- Any abnormal (as determined by a physician) screening laboratory test results
- Any history of neurologic disease (including migraines or seizures)
- Any history of psoriasis (itchy skin rash) or porphyria (rare disturbance of metabolism), since these conditions could get worse after treatment with chloroquine (a medication for treating malaria).
- You have had your spleen removed
- Any past or current infection with HIV, Hepatitis C, or Hepatitis B
- Any use of investigational drugs or vaccines within 1 month before starting the study
- Any allergy to or inability to take the anti-malaria medications used in this study
- Any history of allergic reaction to mosquito bites that required hospitalization
- You must not be pregnant or nursing, or have any plans to become pregnant or breastfeed during the period from now through 3 months after malaria challenge
- Any chronic use of steroids or other medications that affect the immune system in the 6 months before malaria challenge. Inhaled and topical (used on the skin) steroids are allowed.
- You plan to have surgery between enrollment and 3 months after malaria challenge.
- Any active alcohol or drug abuse

 You have any other physical or psychologic condition or laboratory abnormality that the study doctor thinks may increase your risk of having side effects or compromise the results of the study.

#### What are my responsibilities as a participant in this research study?

If you agree to participate in this study, you will be expected to keep all of your study visit appointments. If you cannot make your scheduled appointment, call the WRAIR CTC at 301-319-9660 during operating hours (Monday to Friday 06:00AM to 2:30PM).

#### What happens to the information and specimens collected for this research?

Information and data collected from you for this research will be used to help us determine whether the new batch of malaria parasites act just like the old batch of parasites, and can cause predictable malaria infection in humans.

The blood samples you provide during the study will be used for laboratory tests to assess your safety, to help us diagnose you with malaria and/or confirm your successful treatment, and to compare different methods of malaria diagnosis. In addition, one sample of blood will be taken and mixed with blood from other subjects to make what are known as positive control pools. A positive control pool is an anonymous blood collection known to be infected with malaria that is used to make sure malaria laboratory tests are working properly. Any blood left over after pool creation will be stored, with your permission, for future use in malaria research.

Any information discovered from your data or samples during this trial that may negatively impact your health (for example, if we discover you have high blood pressure or hepatitis) will be shared with you, and if appropriate you will be counselled by a study investigator and referred to a health care provider for further evaluation and care.

After the study is complete, you may request to find out the overall results (how many of the subjects were infected by the new lot of parasites) from the study investigators.

Your data and samples will not have your name or other identifying information about you. Your data and samples will be labeled by a code (such as a number) and may be sent to investigators at WRAIR or other research scientists throughout the country who work with us, without asking for your permission.

No whole genome sequencing will be conducted on your samples in this study. Whole genome sequencing involves the analysis and description of your entire genetic code, or DNA.

Your stored samples will be used for research only and will not be sold. Research using your blood samples may help develop new products in the future that have the potential for commercial profit, but you will not receive payment for such products.

It is your choice as to whether we can use your blood samples for future research. You can still participate in this study regardless of your decision related to blood samples to be used for future malaria research. Future research using the specimens collected from you might include work to develop and evaluate new products to prevent or treat malaria. However, any future use of your samples will not include whole genome sequencing. You will not be informed if and when this future research occurs or what results come from it.

Once the study is complete, your records will be kept in secure storage at WRAIR for a period of at least 2 years. Records will be maintained until it has been deemed no longer necessary to retain them by the study Sponsor (US Army Surgeon General), and then destroyed as per applicable regulations. Any remaining blood specimens will be kept at WRAIR. Storage and destruction of these samples will be as per the applicable facility Standard Operating Procedures (SOPs). These samples, either individually, or in pool form, will be stored for a maximum of 20 years (counting from when the last subject performed the last study visit), unless local rules, regulations or guidelines arise in the interim which require different timeframes or different procedures.

Any future research using your data will require a research protocol and approval by an Institutional Review Board (IRB) (a committee responsible for protecting research participants) or other authorized official responsible for protecting human subjects in research studies. For instance, an IRB reviewed and approved this current study that you are taking part in. The data protections for privacy and confidentiality described in this document will apply to any future use of your stored data and samples.

#### What are the risks if I participate in this research?

If you decide to participate in this study, you should carefully consider the risks, which are described below. While participating in this study, you are not allowed to participate in any other clinical trial. We will share information about new risks with you as the study continues.

#### **Risks of Drawing Blood**

Blood will be drawn from a vein in your arm using a needle. Blood drawing may cause pain and bruising at the site where the blood is drawn. There is also a small possibility that the area from where the blood is drawn may get infected. Redness and swelling around the site where blood is drawn may be a sign of infection. Sometimes people feel lightheaded or even faint when blood is being drawn. There is also a risk of getting anemia from the repeated blood draws.

We do the following to lower the risks:

- Blood is always collected using standard aseptic techniques to prevent infection.
- No more than 30 tablespoonsful (450 mL) of blood will be drawn during any 8week period.

#### **Risks of Getting Mosquito Bites (During Malaria Challenge):**

You might develop redness, mild swelling, and itching on your arm where the mosquitoes bite you. We will have anti-itch cream available if you would like it. There have been very rare reports of severe allergic reactions after mosquito bites. This type of reaction occurs immediately after the bite and can be very serious. You will be observed in the Clinical Trials Center (CTC) for 30 minutes after you are bitten by mosquitoes. The staff of the CTC is trained to recognize allergic reactions and start treatment early. Equipment and medications to treat allergic reactions are available in the CTC and in the room where you will be bitten by mosquitoes. There have been NO reported human cases of HIV, Hepatitis B, or Hepatitis C being transmitted by mosquitoes; however, the blood used to infect the mosquitoes is provided by a blood donor. This blood will be tested for a large panel of blood-borne diseases, to include HIV, Hepatitis B, and Hepatitis C, syphilis, HTLV-1/2, West Nile Virus, and Trypanosoma cruzi (Chagas disease), and only be used if it is found to be negative for all of them. Additionally, there is also a very small risk that the mosquitoes that bite you could give you a disease other than malaria that we have no way of identifying ahead of time. We take several steps to reduce these theoretical risks:

- The mosquitoes used for challenge are hatched and raised in a controlled laboratory and do not feed on any other person before they bite you.
- Blood that is used to feed mosquitoes is obtained from healthy US volunteers
  with normal screening labs. As above, we test all blood that is used to feed
  mosquitoes to make sure that it is negative for Hepatitis B, Hepatitis C, HIV,
  syphilis, West Nile Virus, *Trypanosoma cruzi* (Chagas disease) and Human T
  Lymphotropic Virus (HTLV).

#### **Risks of Getting Malaria**

Infection with the type of malaria mentioned in this study is serious. If treatment is delayed, it may progress to multi-organ failure, seizures, and death. This is why it is so important that you come to each and every clinic visit after the challenge to be monitored and treated as soon as the malaria infection is found. The malaria challenge is considered safe because people are treated as soon as they are found to have a small amount of malaria. Over the past 30 years, both Army and Navy doctors have worked on studies where malaria-infected mosquitoes have bitten more than 1,500 volunteers. All volunteers have recovered from their malaria infections, no volunteers have ever been hospitalized for their infections, and none have ever died of malaria. You are not contagious to others after you develop malaria infection. If you become positive for malaria during this study and complete treatment; malaria symptoms should not recur. If you do not become infected with malaria during the study, it is very unlikely that you will become sick after that. Please contact the CTC staff immediately or tell your personal doctor if you develop symptoms of malaria in the 6 months after the follow up visit. In the extremely unlikely event that malaria does recur we will make sure you receive appropriate evaluation and treatment. To reassure you, no one ever

experimentally infected with this strain of malaria (NF54 clone 3D7) has ever had a recurrence of malaria after completing treatment.

Due to American Red Cross regulations, you will not be allowed to donate blood for 3 years after being exposed to malaria. **Infection with malaria does not protect you from getting malaria if you travel and are exposed to malaria again in the future.** If you travel to a country with malaria later, you still need to take all safety measures to prevent getting malaria such as taking anti-malarial medications.

You should be aware that the medications used to treat malaria in this study may uncommonly produce side effects in individuals taking them. These side effects are discussed further elsewhere in this document.

#### **Risk of Loss of Confidentiality**

If you participate in this study, there is a chance that limited information about you may be released to persons outside of this study, as explained in detail elsewhere in this document.

#### Risks during pregnancy

#### You should not get pregnant or breastfeed while taking part in this study.

Malaria infection during pregnancy is dangerous to both a pregnant woman and her fetus, and can be life-threatening to both. As such, pregnant women are not allowed to participate in this trial for safety reasons.

Malaria infection is not known to be transmitted to infants through breast feeding. However, some medications used to treat malaria can be transmitted to infants through breast milk, and potentially expose those infants to the side effects of those medications. As such, breastfeeding women are not allowed to participate in this trial for safety reasons.

If you are a female who is able to become pregnant and you want to take part in this study, you must agree to consistently use effective birth control (e.g., oral or implanted contraceptives, intrauterine device (IUD), diaphragm with spermicide, abstinence, cervical cap) during the period from the day of screening (today) through 3 months after the malaria challenge. You will also have to take a urine pregnancy test today, and prior to being exposed to malaria. If either of these tests are positive, you will not be allowed to participate in this study.

If during this study you become pregnant or feel you might be pregnant, contact your personal physician and the principal investigator of this study listed in the Contact Information section at the end of this document. If you become pregnant during the study after being exposed to malaria, but before being diagnosed with malaria infection, you will be treated immediately as if you have malaria, with an appropriate drug from those described in the **Treatment of Malaria** section below.

#### **Risks of Heart Disease**

We do not believe the malaria challenge will cause heart disease; however, 3 individuals who took part in malaria challenges in Holland are known to have suffered from heart disease during these studies. None of those events was felt to be caused by the challenge. Instead, the heart disease was felt to be coincidental to the challenge in all 3 cases. The challenge was different than ours and the treatment medications used were not FDA-approved. This is why we need to ask you questions about your health before starting the study and check your heart rate and blood pressure at every visit. For your safety, if you are naturally prone to a moderate or higher risk of getting heart disease, you will not be allowed to participate in the study.

#### **Unknown or Unanticipated Risks**

There may be risks that are not known at this time or that have not been reported yet. If any new risk is reported, the study doctors will let you know as soon as possible.

#### Precautions for volunteers undergoing malaria challenge

Certain antibiotics (medicines that fight infection) can prevent or delay malaria parasites from growing. If your personal physician prescribes an antibiotic for you to be taken any time during the period from 4 weeks before the malaria challenge through the end of the study, you should tell a study physician, before you begin to take it if possible. For safety purposes and study integrity, if the study physician finds that this antibiotic might affect malaria parasites, you may not be allowed to participate in the malaria challenge, or if you are in the study, you may be withdrawn from it.

You should not travel outside the Baltimore/Washington DC area for 28 days after the malaria challenge. If you do have or make travel plans, please let the clinical team know about any travel plans you may have so we can coordinate your visits and give you safety advice.

Participating in this malaria challenge will not protect you from getting malaria in the future. After you complete the study, you should take normal steps to prevent malaria as recommended by your doctors. You will not be able to donate blood at the Red Cross or any other blood collection center, during the study and for 3 years after the malaria challenge.

#### **Treatment for Malaria**

We will treat you with Malarone, which is FDA-approved for treating malaria. If you are allergic to Malarone, or a physician investigator feels that based on your medical history a different medication would be more appropriate, we will treat you with either chloroquine or Coartem, which are also FDA-approved malaria treatment.

The following side effects of Malarone are uncommon and occur in less than 5% of people who take this medication:

- · Abdominal pain, nausea, vomiting
- Temporary elevation of liver function tests.

Version 4, Date: <u>21FEB2019</u>

Headache

If you receive chloroquine for treatment, you may have any of the following side effects:

- Abdominal cramps, loss of appetite, diarrhea, nausea, or vomiting,
- Headache, difficulty sleeping, dizziness, or blurred vision
- Itching
- Tinnitus (ringing in ears) or decreased ability to hear if you already have an existing hearing problem.
- When taken for a long period of time (greater than 1 month), chloroquine can cause permanent eye damage or deafness. Please note that your chloroquine treatment course will last for only 3 days, so it will be highly unlikely that you would develop eye damage or deafness from the medication.

If you receive Coartem for treatment, you may have the following side effects:

- Fever, chills, headache, dizziness, weakness, difficulty sleeping
- Loss of appetite, abdominal pain, nausea, vomiting
- Muscle aches, joint aches
- Cough

#### How will my privacy and data confidentiality be protected?

We will take measures to protect your privacy. Even with these measures, we can never fully guarantee your privacy will be protected. We will try our best to protect your privacy by doing the following:

- Your name and any identifiable information (for example, your address or social security number) will be removed from study files and your lab samples and be replaced with an identification code that consists of numbers and letters. Different codes may be used for you during the course of the study. Only the study investigators, study coordinators, research monitor and representatives from certain agencies (described below) will be allowed to know which codes belong to you, and to have access to your study information.
- Your study files will be kept in a safe, secure storage area at the WRAIR Clinical Trials Center for the duration of the study.

While we will do our best to protect your information there are some cases where we cannot guarantee complete confidentiality.

We may report medical information and lab results to authorities, to prevent serious harm of yourself or others.

• We are required to report information regarding certain infectious diseases (like HIV or AIDS and viral hepatitis) to the local health department. If your blood tests show that you have one of these infections, we will report this information to the health department, and they may need to interview you to get more information. This may cause you some distress, and could affect your personal and professional relationships. We will provide trained counselling to discuss test results and refer you for further care as required.

- For volunteers who are in the military, information bearing on your health may
  be required to be reported to appropriate medical or command authorities.
  This may include information bearing on your safety, the safety of others, or
  your ability to perform your duties (for example, evidence of suicidal or
  homicidal behavior). It also may include information that indicates possible
  substance abuse or other potential criminal activity under the Uniform Code of
  Military Justice.
- Representatives from the following agencies may have access to review research records as part of their responsibility to protect humans in research and oversee the quality of the research efforts. As government agencies, they must also maintain confidentiality of your records within the limits of the law.
  - The Study Sponsor, US Army Surgeon General
  - The WRAIR Institutional Review Board (IRB)
  - The Naval Medical Research Center (NMRC) Institutional Review Board (IRB)
  - U.S. Army Medical Research and Materiel Command (USAMRMC)
  - The US Food and Drug Administration

Please remember that even though we are doing our best to protect your information, we can never fully guarantee confidentiality of all study information.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### Will I be paid to take part in this research study?

Yes, for your participation, you will receive compensation. Compensation will be provided at each visit for completed study procedures. If you participate in the study, you will be compensated as follows:

- Screening visit: \$50 per completed visit
- Malaria challenge (1 visit): \$275

 Post challenge Pre-hotel clinic visits (9 visits): \$100 per completed visit. For days with multiple visits, there will be a maximum compensation of \$100 per day, and payment may be bundled and provided after completion of the final visit of the day.

- Hotel phase (up to 10 nights after the malaria challenge): \$100 per day for a
  total of \$1000 regardless of when you develop malaria provided that you
  attend all of the required hotel stay daily study visits, including the follow-up
  visits after malaria treatment is started. If you fail to attend all of the required
  visits, your payment for this portion will be reduced to reflect your actual
  participation.
- (If needed) Post-hotel phase follow-up visits with a blood draw to complete treatment and/or confirm parasite clearance (Up to approximately 3 visits): \$100 per completed visit. For days with multiple visits, there will be a maximum compensation of \$100 per day, and payment may be bundled and provided after completion of the final visit of the day.
- Unscheduled visit requiring a blood draw: \$50 per visit
- Final Study Visit with blood draw: \$100+ (if eligible) \$250 bonus for completion of all required study visits.

If you are a federal employee (military or civilian), participating while on-duty, your compensation will be \$50 per visit with a blood draw. However, if your visit with a blood draw occurs during off-duty hours or while you are on leave, your compensation will be the same as that for non-federal personnel.

In order to participate on- or off-duty, active duty military volunteers will require approval from their supervisor through division director using the Statement of Supervisor's Approval, which will be provided to you.

The maximum possible compensation for a volunteer who attends all study visits amounts to approximately \$2,875.00. The maximum possible compensation for an **on-duty** federal employee amounts to approximately \$1250. By law, we must report compensation totaling over \$600 provided to any volunteer in single calendar year to the Internal Revenue Service. Please note that we will not provide extra money to pay for costs you may have from being in this study, such as the cost of transportation to and from the study site or child care costs.

If you choose to leave or are removed from the study by the Principal Investigator prior to its completion, you will still be eligible for the compensation related to all study visits and procedures that you have successfully completed up until that point. If you do not complete all required study visits, you will not be eligible for the end of study bonus.

Other than medical care that may be provided and any other payment specifically stated in this informed consent, there is no other compensation available for your participation in this research study; however, you should also understand that this is not a waiver or release of your legal rights.

#### Are there costs for participating in the research?

There is no cost to you to participate in the study. You will not have to pay for medical visits, physical examinations, blood tests, medical procedures, or hospitalizations that occur as a result of this study. However, we will not pay for any transportation or childcare costs.

## Are there disclosures of financial interests or other personal arrangements from the research team?

The Principal Investigator and members of the research team have no financial interests or personal arrangements related to this trial to disclose at this time.

#### What happens if I am injured as a result of this research?

If you are injured because of your participation in this research and you are a Department of Defense (DoD) healthcare beneficiary (e.g. active duty in the military, military spouse or dependent, retiree), you are entitled to medical care for your injury within the DoD healthcare system, as long as you remain a DoD healthcare beneficiary. This care includes but is not limited to free medical care at DoD hospitals or clinics.

If you are injured because of your participation in this research and you are not a DoD healthcare beneficiary, you are entitled to medical care for your injury at an Army hospital or clinic; medical care charges for care at an Army hospital or clinic will be waived for your research-related injury. You are also entitled to care for your injury at other DoD (non-Army) hospitals, but such care for your injury at other DoD (non-Army) hospitals or clinics may be time-limited, and your insurance may be billed. It cannot be determined in advance which Army or DoD hospital or clinic will provide care. If you obtain care for research-related injuries outside of an Army or DoD hospital or clinic, you or your insurance will be responsible for medical expenses.

Transportation to and from hospitals or clinics will not be provided. No reimbursement is available if you incur medical expenses to treat research-related injuries. No compensation is available for research-related injuries. You are not waiving any legal rights.

If you believe that you have sustained a research-related injury, please contact the PI, James E. Moon, MD, or the WRAIR Clinical Trials Centers, whose contact information is given at the top of this document. In addition, an emergency contact card will be provided to you with numbers to contact at any time.

#### What happens if I withdraw from this research?

**PARTICIPATION IN THIS STUDY IS VOLUNTARY.** You may decide not to take part in this study. You can withdraw from (leave) this study at any time and for any reason without penalty or loss of benefits to which you are otherwise entitled. However, for your safety, we may need to continue to monitor or provide treatment to you. If you withdraw

Version <u>4</u>, Date: <u>21FEB2019</u>

following the challenge you will be asked to complete follow-up visits, diagnostic tests for malaria, treatment, and safety blood work to ensure your safety.

If you decide to leave the study, we ask you to contact a study investigator or the CTC staff. The information you provided prior to withdrawal will be stored and treated in the same way as for other volunteers. Any data and specimens collected prior to your withdrawal will be used by the study in the same ways as for other volunteers. No more payments will be made to you after the final blood work. The quality of the medical care you receive will not be affected by your decision to withdraw from the study.

The principal investigator, James Moon, MD, may decide not to allow you to continue participating in this study under the following conditions:

- If you develop a medical condition that would make it unsafe for you or others
  if you were to continue participating, or that would interfere with the study
  results
- If other situations or conditions arise that would make participation harmful to your own health,
- If you fail to comply with the procedures as outlined in this form.
- If the study ends for any reason.
- If the investigator believes that it is in your best interest.

You should also know that the WRAIR Institutional Review Board (IRB), and the US Army Medical Research and Materiel Command (USAMRMC) can end this study at any time. If the study ends, or your participation ends, you may be asked to complete follow-up visits and/or medication for your safety.

We will tell you if we discover any significant or new information during the study that may affect your health and willingness to continue participation.

#### Who can I contact if I have questions about my rights as a research participant?

If you have questions about your rights as a research volunteer in this study, you may contact the Human Subjects Protection Branch, Walter Reed Army Institute of Research 503 Robert Grant Avenue, Silver Spring, MD 20910, phone number 301-319-9940 and email usarmy.detrick.medcom-wrair.mbx.hspb@mail.mil.

#### What is the volunteer registry?

It is the policy of the U.S. Army Medical Research and Materiel Command (USAMRMC) that data sheets are to be completed on all volunteers participating in research for entry into this Command's Volunteer Registry Data Base. The information to be entered into this confidential data base includes your name, address, Social Security number, study name and dates. The intent of the data base is two-fold: first, to readily answer questions concerning an individual's participation in research sponsored by USAMRMC; and second, to ensure that the USAMRMC can exercise its obligation to ensure research volunteers are adequately warned (duty to warn) of risks and to provide new information as it becomes available. The information will be stored at USAMRMC for a

minimum of 75 years. The Volunteer Registry Data Base is separate from and not linked to the treatment protocol database.

#### Consent

If there is any portion of this document that you do not understand, ask the investigator before signing the form. Signing this form means that you consent to participate in this research, at this time.

Please initial the sentences that reflect your choices, and then sign below:

A signed and dated copy of this document will be given to you.

| riodoo iintidi tiio oontonooo tiidt ronoot your or | ioroco, una trion orgin borowi |
|---|---|
| (initials) I do not authorize the storage of my biological specimens for use in future malaria research studies. | |
| (initials) I authorize the storage of my biological specimens for use in future malaria research studies. | |
| SIGNATURE OF PARTICIPANT | |
| Printed Name of Participant | - |
| Signature of Participant | - Date |
| Permanent Address of Participant | |

#### SIGNATURE OF INDIVIDUAL ADMINISTERING CONSENT

(Can only be signed by an investigator or staff approved to administer consent)

**WRAIR #\_2572**Version 4, Date: 21FEB2019

| Printed Name of Administering Individual | |
|------------------------------------------|----------|
| Signature of Administering Individual | <br>Date |